CLINICAL TRIAL: NCT03981484
Title: REPlaCE- Randomized Trial Evaluating the Use of Prothrombin Complex concEntrate to Improve Survival in Patients With Traumatic Coagulopathy
Acronym: REPLaCE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bellal A. Joseph, MD, FACS (Other)
Responsible Party: Sponsor-Investigator, Bellal A. Joseph, MD, FACS, Chief of the Division of Trauma, Acute Care, Burn, and Emergency Surgery, University of Arizona
Organization: University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00001
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Coagulopathy; Hemorrhage
MeSH Terms: conditions — Hemostatic Disorders; Hemorrhage | interventions — Factor IX

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCC (Experimental): single dose of 4-Factor PCC in addition to standard resuscitation methods
  Interventions: Biological: Prothrombin Complex Concentrate
- Standard of Care (Active Comparator): standard resuscitation methods only
  Interventions: Biological: Whole Blood, Plasma, Packed Red Blood Cells

INTERVENTIONS:
Biological: Prothrombin Complex Concentrate — single dose of 25 IU/kg of 4-PCC at time of enrollment
  Arms: PCC
Biological: Whole Blood, Plasma, Packed Red Blood Cells — site's standard resuscitation protocol
  Arms: Standard of Care

SUMMARY:
Uncontrolled hemorrhage continues to be a significant source of mortality for trauma patients. Their condition is further complicated by Trauma Induced Coagulopathy (TIC), which makes it more difficult to control bleeding due to coagulation factor deficiency. Prothrombin Complex Concentrate (PCC) is thought to be a promising treatment option. This phase II clinical trial evaluates the use of 4-Factor PCC in addition to standard resuscitation methods compared to standard resuscitation methods alone in patients with TIC. Patients will be randomized at a 1:1 ratio. The primary endpoint of this trial will be 30 day mortality.

ELIGIBILITY:
Inclusion Criteria:

1. ≥15 years old
2. anticipate giving 4+ units based on Revised Assessment of Bleeding and Transfusion score ≥ 2

Exclusion Criteria:

1. Cardiopulmonary Resuscitation > 5 minutes
2. Penetrating cranial injury or exposed brain matter
3. Anticoagulation treatment
4. Transfer patients
5. Known pregnancy
6. Prisoners

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
24 Hour Mortality | 24 hours after enrollment
  Assess if patient is alive at 24 hours post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bellal Joseph, MD, Principal Investigator — University of Arizona

IPD SHARING:
Plan to Share IPD: No